CLINICAL TRIAL: NCT04632745
Title: A Prospective Randomized Evaluation of Splinting and Casting for Distal Radius Fractures in the Elderly
Brief Title: A Study Evaluating Splinting and Casting for Distal Radius Fractures in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JMAT20D.390
Record Dates: First submitted 2020-10-29; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cast Group (Other): participant with distal radius fracture will be treated with short arm fiberglass cast
  Interventions: Other: Wrist Rehabilitation
- Splint Group (Other): participant with distal radius fracture will be treated with short arm velcro wrist splint
  Interventions: Other: Wrist Rehabilitation

INTERVENTIONS:
Other: Wrist Rehabilitation — participants will undergo immobilization for the first 6 weeks of treatment

SUMMARY:
Distal radial fractures are the most common fracture of the upper extremity in adults, with a higher incidence in those 65 years of age or older. In 2009, Karl et al demonstrated that there are 25.42 distal radial fractures in this age group per 10,000 person-years in the US. Despite the frequency of distal radius fractures, there is still debate over the best method of treatment. In contrast to younger patients, patients who are 65 years or older appear to have acceptable functional outcomes and treatment satisfaction regardless of the presence of malalignment on radiographic imaging.Therefore, nonsurgical management has been shown to be a viable treatment option.

The purpose of this study is to compare non-operative treatment with a removable splint versus a short arm cast for distal radial fractures in patients who are 65 years of age or older who are indicated for non-operative fracture treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 65 years old with isolated distal radius fracture amenable to non-operative treatment

Exclusion Criteria:

* Patients younger than 65 years old
* Open fractures (Gustilo Grade 2 or 3)
* Pathologic fractures
* Multiple fractures in the upper or lower extremities
* Fracture indicated for surgical repair of the distal radius for any reason
* Lack of health insurance
* Inability to provide consent to the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Fracture treatment outcome | 6 weeks
  The rate of successful outcomes of participants who are treated for a distal radius fracture nonsurgically by splinting compared to participants who are treated by casting

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States